CLINICAL TRIAL: NCT05782907
Title: A Phase 3 Multicenter Study to Evaluate Efficacy, Safety, and Pharmacokinetics of Upadacitinib With Open-Label Induction, Randomized, Double-Blind Maintenance and Open-Label Long-Term Extension in Pediatric Subjects With Moderately to Severely Active Ulcerative Colitis and Inadequate Response, Intolerance, or Medical Contraindications to Corticosteroids, Immunosuppressants, and/or Biologic Therapy
Brief Title: Study to Assess Adverse Events, Change in Disease Activity, and How Oral Upadacitinib Moves Through the Body of Pediatric Participants With Moderately to Severely Active Ulcerative Colitis.
Acronym: U-ASTOUND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-658; 2022-501788-41-00 (Other: EU CT)
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
Keywords: Upadacitinib; RINVOQ; Ulcerative Colitis; UC; Corticosteroids; Immunosuppressants; Biologic Therapy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Period 1- Open Label Induction Phase (Experimental): All participants in open label induction phase of Period 1 will receive upadacitinib Dose A for 8 weeks based on body weight.
  Interventions: Drug: Upadacitinib
- Period 1- Double Blind Maintenance Phase (Experimental): Clinical responders at the end of open label induction phase of Period 1 will be randomly assigned to receive either upadacitinib Dose B or Dose C for 44 weeks based on body weight.
  Interventions: Drug: Upadacitinib
- Period 2- Open Label Long Term Extension Phase Arm A (Experimental): Clinical non-responders outside of US after Period 1 induction phase will receive upadacitinib Dose A daily for 8 week extended induction phase in open label long term extension (OLE) Period 2. Clinical responders from extended induction phase in OLE will receive upadacitinib Dose B daily for up to 252 weeks in OLE period 2.
  Interventions: Drug: Upadacitinib
- Period 2- Open Label Long Term Extension Phase Arm B (Experimental): Clinical non-responders in US after Period 1 induction phase or clinical responders with loss of response during maintenance phase will receive upadacitinib Dose B daily for up to 260 weeks in OLE Period 2.
  Interventions: Drug: Upadacitinib
- Period 2- Long Term Extension Phase Arm C (Experimental): Clinical responders who complete Period 1 through Week 52 will receive upadacitinib Dose C daily for up to 260 weeks in OLE Period 2.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Oral Solution/ Tablets
  Other Names: RINVOQ

SUMMARY:
Ulcerative colitis (UC) is a type of inflammatory bowel disease that causes inflammation and bleeding from the lining of the rectum and colon (large intestine). This study will assess how safe and effective Upadacitinib is in treating pediatric participants with UC. Adverse events and change in disease activity will be assessed.

Upadacitinib (RINVOQ) is a drug approved in adults for moderate- to severely active UC and is being developed for moderate- to severely active UC in pediatric participants. This study is conducted in 2 periods: Period 1 is comprised of two phases: an 8-week open-label induction phase which means that the study doctor and patients know that participants will receive UPA Dose-A (or the adult equivalent based on body weight) followed by a 44-week double-blind maintenance phase meaning that neither the participants nor the study doctors will know which dose of upadacitinib will be given(UPA Dose B or Dose C). Period 2 is a 260 week open-label extension (OLE) of Period 1. Approximately 110 pediatric participants with moderate to severely active UC will be enrolled at up to 100 sites worldwide.

Participants will receive upadacitinib oral tablets once daily or oral solution twice daily at approximately the same time each day, with or without food. Participants will be followed up for 30 days after each phase (i.e. after induction, maintenance, OLE) and only if a participant doesn't continue into the next phase.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Active UC with an AMS of 5 to 9 points and endoscopic subscore of 2 to 3.
* Demonstrate an inadequate response, loss of response, intolerance, or medical contraindications to corticosteroids, immunosuppressants, and/or biologic therapy.

Exclusion Criteria:

* Partcipants with previous exposure to JAK inhibitors (e.g., tofacitinib, baricitinib, filgotinib, upadacitinib).
* Females who are pregnant, breastfeeding, or considering becoming pregnant during the study and for approximately 30 days after the last dose of study drug.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Adapted Mayo score (AMS) Clinical Remission (Period 1) | Week 8
  The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The AMS is a composite of the following subscores: stool frequency subscore (SFS), rectal bleeding subscore (RBS) and endoscopy subscore (MES). AMS ranges from 0 to 9 where higher scores represent more severe disease. Clinical remission is defined as an AMS < or = 2, with SFS < or = 1 and not higher than baseline, RBS of 0, and MES < or = 1.
Percentage of Participants Achieving AMS Clinical Remission Among Week 8 Responders per AMS (Period 1) | Week 52
  The Mayo score is a tool designed to measure disease activity for ulcerative colitis. AMS ranges from 0 to 9 where higher scores represent more severe disease. Clinical remission is defined as an AMS ≤ 2, with SFS ≤ 1 and not higher than Baseline, RBS of 0, and MES ≤ 1.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Endoscopic Improvement (Period 1) | Week 8
  Endoscopic Improvement is defined as MES < or = 1.
Percentage of Participants Achieving Partial Mayo Score (PMS) Clinical Remission (Period 1) | Week 8
  The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The PMS is a composite of the following subscores: SFS, RBS and physician's global assessment (PGA). The PMS ranges from 0 to 9 with higher scores representing more severe disease. PMS clinical remission is defined as a PMS < or = 2 and no individual subscore > 1.
Percentage of Participants Achieving AMS Clinical Response (Period 1) | Week 8
  The adapted mayo score (AMS) is a composite of the following subscores: SFS, RBS and MES. AMS clinical response is defined as decrease in AMS by > or = 2 points and > or = 30% from baseline with a decrease in RBS of > or = 1 or an absolute RBS of 0 or 1.
Percentage of Participants Achieving Endoscopic Improvement Among Week 8 Responders per AMS (Period 1) | Week 52
  Endoscopic Improvement is defined as MES of < or = 1. The AMS is a composite of the following subscores: SFS, RBS and MES.
Percentage of Participants Achieving PMS Clinical Remission Among Week 8 Responders per AMS (Period 1) | Week 52
  The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The PMS ranges from 0 to 9 with higher scores representing more severe disease. PMS clinical remission is defined as a PMS < or = 2 and no individual subscore > 1. The AMS is a composite of the following subscores: SFS, RBS and MES.
Percentage of Participants Achieving AMS Clinical Response Among Week 8 Responders per AMS (Period 1) | Week 52
  The AMS is a composite of the following subscores: SFS, RBS and MES. AMS clinical response is defined as decrease in AMS by > or = 2 points and > or = 30% from baseline with a decrease in RBS of > or = 1 or an absolute RBS of 0 or 1.
Percentage of Participants Achieving PMS Clinical Response Among Week 8 Clinical Responders per AMS (Period 1) | Week 52
  The AMS is a composite of the following subscores: SFS, RBS and endoscopy MES. PMS clinical response is defined as decrease in PMS by > or = 2 points and > or = 30% from baseline with a decrease in RBS > or = 1 or an absolute RBS of 0 or 1.
Percentage of Participants Achieving Corticosteroid-Free AMS Clinical Remission Among Week 8 Responders per AMS (Period 1) | Week 52
  Corticosteroid-free AMS clinical remission is defined as being in AMS clinical remission and free of corticosteroids for >= 90 days immediately preceeding the timepoint of endpoint assessment. The AMS is a composite of the following subscores: SFS, RBS and MES.
Percentage of Participants Achieving AMS Clinical Remission Among Week 8 Remitters per AMS (Period 1) | Week 52
  The AMS is a composite of the following subscores: SFS, RBS and MES. Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease. Clinical remission is defined as an AMS < or = 2, with SFS < or = 1 and not higher than baseline, RBS of 0, and MES < or = 1.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (89):
- United States (20):
  - Phoenix Children's Hospital /ID# 250135, Phoenix, Arizona
  - Arkansas Children's Hospital /ID# 250106, Little Rock, Arkansas
  - Kindred Medical Institute - Corona /ID# 255484, Corona, California
  - UCSF Benioff Children's Hospital - Oakland /ID# 255067, Oakland, California
  - Lucile Packard Children's Hospital /ID# 258430, Palo Alto, California
  - Children's Hospital Colorado - Aurora /ID# 250110, Aurora, Colorado
  - Nemours/Alfred duPont Hospital for Children /ID# 255483, Wilmington, Delaware
  - Childrens Healthcare of Atlanta - Center for Advanced Pediatrics /ID# 255069, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago /ID# 254505, Chicago, Illinois
  - OSF St. Francis Medical Center /ID# 256968, Peoria, Illinois
  - Massachusetts General Hospital /ID# 250142, Boston, Massachusetts
  - Boston Children's Hospital /ID# 250108, Boston, Massachusetts
  - NYU Langone Hospital - Long Island /ID# 250136, Mineola, New York
  - The Mount Sinai Hospital /ID# 250141, New York, New York
  - Univ NC Chapel Hill /ID# 254541, Chapel Hill, North Carolina
  - Levine Children's Hospital /ID# 250131, Charlotte, North Carolina
  - UH Cleveland Medical Center /ID# 250134, Cleveland, Ohio
  - Children's Hospital of Philadelphia - Main /ID# 258773, Philadelphia, Pennsylvania
  - Children's Specialty Group /ID# 256966, Norfolk, Virginia
  - University of Wisconsin - Madison /ID# 250632, Madison, Wisconsin
- Australia (4):
  - Children's Hospital at Westmead /ID# 255556, Westmead, New South Wales
  - Queensland Children's Hospital /ID# 261032, South Brisbane, Queensland
  - Monash Health - Monash Medical Centre /ID# 254726, Clayton, Victoria
  - Perth Children'S Hospital /ID# 254727, Perth, Western Australia
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen /ID# 251184, Edegem, Antwerpen
  - Universitair Ziekenhuis Leuven /ID# 251185, Leuven, Vlaams-Brabant
- Brazil (3):
  - Hospital Pequeno Príncipe /ID# 251911, Curitiba, Paraná
  - Hospital e Maternidade Celso Pierro - PUC-Campinas /ID# 251912, Campinas, São Paulo
  - Rocco & Nazato Servicos Medicos /ID# 251910, São Paulo, São Paulo
- Bulgaria (3):
  - UMHAT Sveti Georgi /ID# 251949, Plovdiv
  - Specialized Hospital For Active Treatment Of Children Diseases Prof. Ivan Mitev /ID# 251285, Sofia
  - UMHAT Multiprofile Hospital for Active Treatment Sveta Marina /ID# 251948, Varna
- Canada (5):
  - Alberta Health Services /ID# 252088, Edmonton, Alberta
  - South Edmonton Gastroenterology /ID# 276669, Edmonton, Alberta
  - BC Children's Hospital /ID# 250947, Vancouver, British Columbia
  - IWK Health Center /ID# 250943, Halifax, Nova Scotia
  - Hospital for Sick Children /ID# 250945, Toronto, Ontario
- Czechia (2):
  - Fakultní Nemocnice Plzeň-Lochotín /ID# 253284, Pilsen, Plzen-jih
  - Fakultní nemocnice v Motole /ID# 251955, Prague, Praha 5
- France (5):
  - CHU Bordeaux - Hopital Pellegrin /ID# 253182, Bordeaux, Nouvelle-Aquitaine
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant /ID# 251502, Bron, Rhone
  - AP-HP - Hopital Necker /ID# 251658, Paris
  - Hopitaux de Paris (AP-HP) - Hopital Robert Debre - CHU /ID# 252069, Paris
  - CHU Toulouse - Hopital Paule de Viguier /ID# 252070, Toulouse
- Germany (4):
  - Dr. von Haunerschen Kinderspital /ID# 251440, Munich, Bavaria
  - Universitaetsklinikum Muenster /ID# 256763, Münster, North Rhine-Westphalia
  - Klinikum St. Georg gGmbH /ID# 262481, Leipzig, Saxony
  - Charite Universitaetsmedizin Berlin Campus Virchow-Klinikum /ID# 251434, Berlin
- Greece (2):
  - Agia Sofia Hospital /ID# 250697, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 250696, Heraklion, Crete
- Hungary (2):
  - Debreceni Egyetem-Klinikai Kozpont /ID# 251835, Debrecen, Hajdú-Bihar
  - Semmelweis Egyetem /ID# 251083, Budapest
- Israel (2):
  - Schneider Children's Medical Center /ID# 254833, Petah Tikva, Central District
  - Shaare Zedek Medical Center /ID# 254832, Jerusalem, Jerusalem
- Italy (3):
  - Azienda Ospedaliero Universitaria Meyer /ID# 251624, Florence, Firenze
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 251625, Rome, Roma
  - Ospedale Maggiore Carlo Alberto Pizzardi /ID# 251626, Bologna
- Japan (10):
  - Tsujinaka Hospital - Kashiwanoha /ID# 251930, Kashiwa-shi, Chiba
  - Kurume University Hospital /ID# 251927, Kurume-shi, Fukuoka
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 251928, Sapporo, Hokkaido
  - Miyagi Children's Hospital /ID# 251931, Sendai, Miyagi
  - Osaka Women's and Children's Hospital /ID# 252397, Izumi-Shi, Osaka
  - Osaka General Medical Center /ID# 253678, Osaka, Osaka
  - Saitama Children's Medical Center /ID# 252362, Saitama-shi, Saitama
  - Institute of Science Tokyo Hospital /ID# 251929, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Children's Medical Center /ID# 252477, Fuchu-shi, Tokyo
  - National Center For Child Health And Development /ID# 251926, Setagaya City, Tokyo
- Servicios de Oncologia Medica Integral SA de CV /ID# 252974, San Pedro Garza García, Nuevo León, Mexico
- Netherlands (2):
  - Amsterdam UMC, locatie AMC /ID# 250845, Amsterdam, North Holland
  - Universitair Medisch Centrum Groningen /ID# 252003, Groningen
- New Zealand (2):
  - Christchurch Hospital. /ID# 254703, Christchurch, Canterbury
  - Starship Child Health /ID# 254702, Auckland
- Poland (2):
  - Gastromed Sp. z o.o /ID# 251290, Torun, Kuyavian-Pomeranian Voivodeship
  - Instytut Pomnik - Centrum Zdrowia Dziecka /ID# 251289, Warsaw, Masovian Voivodeship
- Clinical Research Puerto Rico /ID# 266477, San Juan, Puerto Rico
- South Korea (3):
  - Seoul National University Hospital /ID# 252024, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 252023, Seoul, Seoul Teugbyeolsi
  - Kyungpook National University Chilgok Hospital /ID# 252663, Daegu
- Spain (4):
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 252105, Ferrol, A Coruna
  - Hospital Sant Joan de Deu /ID# 251194, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Vall de Hebron /ID# 252104, Barcelona
  - Hospital Regional Universitario de Malaga /ID# 251193, Málaga
- Taiwan (2):
  - National Taiwan University Hospital /ID# 251650, Taipei City, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 251654, Taoyuan
- United Kingdom (5):
  - Sheffield Children's Hospital NHS Foundation Trust /ID# 251600, Sheffield, England
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 251917, London, Greater London
  - Great Ormond Street Children's Hospital /ID# 252126, London, Greater London
  - University Hospital Southampton NHS Foundation Trust /ID# 252097, Southampton, Hampshire
  - Birmingham Women's and Children's NHS Foundation Trust /ID# 253072, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.abbvieclinicaltrials.com/study/?id=M14-658